CLINICAL TRIAL: NCT03552328
Title: Effects of a Pilot Volunteer-based Lunch Program on Feelings of Loneliness in Elders: a Randomized Control Trial
Brief Title: Effects of a Volunteer-based Lunch Program on Feelings of Loneliness in Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: The Arnold P. Gold Foundation (Other)
Responsible Party: Principal Investigator, Brennan Ninesling, Medical Student, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00034170
Record Dates: First submitted 2018-05-26; First posted 2018-06-11 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Aged; Loneliness; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Lunch

STUDY DESIGN:
Intervention Model Description: Eligible and consenting participants are randomized to one of the two study groups in a 1:1 allocation ratio. A block-stratified method using the computer will be used for generation of randomization sequence. The block size will be random.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization sequence will be implemented centrally with one of the co-investigator (Ambuj Kumar) who is off site will retain the list. Once a participant is identified the primary investigator will call the off-site co-investigator for assignment. Given that the co-investigator is not on site will ensure adequate allocation concealment.
  Also, since the outcome data will be collected using a questionnaire, the possibility of interpretation does not exist. Data analysts will not be informed of the subject assignment and the coding for participant will be as group 1 or 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Seniors receiving daily meals from Meals on Wheels. Intervention: Lunch with Medical Student.
  Interventions: Other: Lunch with Medical Student
- Control (Placebo Comparator): Seniors receiving daily meals from Meals on Wheels
  Interventions: Other: Control

INTERVENTIONS:
Other: Lunch with Medical Student — Each student will bring provided lunches once a week to their elder participant's residence, and they will share lunch together for an hour once a week for six weeks. Students will enroll as Meals on Wheels volunteers and participate in the Meals on Wheels pre-program training. On the day of their scheduled lunch, students will first arrive at the Meals on Wheels designated meal-drop location and pick up two lunches, one for them and one for their assigned elder. They will then drive to their assigned elder's residence and eat lunch with them for one hour.
  Arms: Intervention
Other: Control — Students will not bring provided lunches to an elder participant's residence. The elder participants in this arm will simply continue receiving daily meals from Meals on Wheels with no accompanying student.
  Arms: Control

SUMMARY:
Background: There is a need for stronger community involvement with the elderly, specifically those with feelings of loneliness. Large proportions of elders in previous studies reported feelings of loneliness, and loneliness at advanced ages is a growing trend seen within the last thirty years despite advances in technology and social media. We propose a randomized control trial to determine the effectiveness of a volunteer-based lunch program on decreasing feelings of loneliness in elderly participants.

Methods: Lonely elders in the community will be identified and matched with a trained medical student. Each student will bring provided lunches once a week to their elder participant's residence, and they will share lunch together for an hour once a week for six weeks. Enrollees are eligible for the study if they are over 60 years of age, speak English, have feelings of loneliness on the three-item scale, and display no cognitive impairment. The participants will be assessed pre and post intervention using the R-UCLA scale for loneliness, PHQ-9 for depressive symptoms, and GAD-7 for feelings of anxiety. Participant satisfaction will be assessed using Likert items as well as open-ended questions. Intervention group responses will be compared to responses of participants that did not receive the lunch meeting intervention.

Discussion: Success of such a companion lunch program would provide an effective route to combat loneliness in the elderly.

DETAILED DESCRIPTION:
Since the 1960's, the elderly population in the United States has grown steadily. By 2030, one in three people in the U.S. will be over the age of 65. In addition to being at a greater risk for chronic disease, the elderly are also more vulnerable to being socially isolated and lonely. Simply living alone does not appear to be a significant predictor of loneliness, as the elderly could still have a strong support network while living alone, but prevalence data suggests that one in three adults over the age of 65 are lonely. Furthermore, the oldest of the elderly seem to be the loneliest. Dykstra et al. in a 2009 study estimate 40 to 50 percent of those aged 80 or older to be lonely.

Loneliness has been previously defined as the difference between desired and actual relationships, and there is a distinction between loneliness and social isolation. While being considered socially isolated is due to lack of social contact, loneliness is assessed by perceptions of social isolation. Feelings of disconnect, isolation, and not belonging are much more indicative of loneliness than simple aloneness and lack of social contact. Not having a support network or anyone to confide in can lead to feelings of social isolation, and despite advances in technology and the development of social media, feelings of loneliness have increased in the past thirty years. The proportion of Americans who said they had no one to talk to about important matters increased from 10% in 1985 to 25% in 2004. This is an alarming trend because social support has been consistently shown to increase the likelihood of survival. In a meta-analytic review from 2009, participants with strong social relationships and support were found to have a 50 percent increased likelihood of survival. Additionally, a 2013 study found that mortality rates were significantly higher among socially isolated and lonely elders. Loneliness has a profound effect on our healthcare system and has been linked to a higher degree of healthcare utilization. In a Swedish study from 2014, researchers found that lonely elders use more outpatient services than non-lonely elders. In 2015, Gerst et al. found that the large proportion of elders over 60 years old that reported feelings of loneliness had a significantly higher physician visit rate.

There is a demonstrated need for intervention in this lonely, elderly population, with significant public health implications. A randomized control trial from 1999 implementing a visitor volunteer program for the elderly showed that strong community involvement increased the participants' feelings of worth, social integration, and life satisfaction. More recently, a local food delivery project in Tampa showed that weekly food delivery to an at-risk elderly population decreased participants' feelings of loneliness and increased their measured well-being over the course of two months. While both pilot programs had short evaluation periods, they demonstrated the effectiveness of volunteer-based community involvement. Combining a visitor volunteer program with a food delivery service could serve to effectively combat the elderly community's feelings of loneliness and social isolation.

A local food delivery project in Tampa showed that weekly food delivery to an at-risk elderly population decreased participants' feelings of loneliness and increased their measured well-being over the course of two months. Even though it demonstrated the effectiveness of volunteer-based community involvement, the project was constructed as a pretest-posttest, descriptive study using convenience sampling, and feelings of loneliness were evaluated as a secondary objective using a three-item loneliness screener. In our study, we plan to measure the effects of adding a volunteer visitor to the lunch program; that is, to see if eating meals with a medical student can decrease feelings of loneliness when compared with simply receiving meals through Meals on Wheels. Our study is designed as a randomized control trial in which seniors will be randomly assigned to two groups: paired with a medical student for lunch or not paired with a medical student while still receiving meals.

ELIGIBILITY:
Inclusion Criteria:

* Enrollees are eligible for the study if they speak English, have feelings of loneliness on the three-item scale, are able to give written consent, and answer surveys.

Exclusion Criteria:

* Elders who are unable to give informed consent or complete trial documentation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-02-17 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Revised-UCLA (R-UCLA) Scale | Survey will be administered on both study groups twice; once before and once after the six-week period.
  Investigators will measure change from baseline feelings of loneliness in elderly participants. Responses are scored from 20 (minimum) to 80 (maximum). Only total scores are reported. Lower values represent a better outcome, i.e. less feelings of loneliness.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Survey will be administered on both study groups twice; once before and once after the six-week period.
  We will measure change from baseline feelings of depression in elderly participants. Responses are scored from 0 (minimum) to 27 (maximum). Only total scores are reported. Lower values represent a better outcome, i.e. less feelings of depression.
Generalized Anxiety Disorder 7-item (GAD-7) Scale | Survey will be administered on both study groups twice; once before and once after the six-week period.
  We will measure change from baseline feelings of anxiety in elderly participants. Responses are scored from 0 (minimum) to 21 (maximum). Only total scores are reported. Lower values represent a better outcome, i.e. less feelings of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Guerra, MD, MPH, Study Director — Associate Professor, USF College of Medicine Internal Medicine
Locations (1):
- Morsani College of Medicine, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We will ensure that all data collected during the trial is handled confidentially and accessed only by members of the team. We will store participants' details on a secure database. We will assign participants an individual specific trial number and we will anonymize their details.

REFERENCES:
- [Background] Lawson, V. and K. Kinsella, Aging in the United States: Past, present, and future. 1996, International Programs Center, Population Division, US Bureau of the Census, Washington, DC.
- [Background] Perissinotto CM, Stijacic Cenzer I, Covinsky KE. Loneliness in older persons: a predictor of functional decline and death. Arch Intern Med. 2012 Jul 23;172(14):1078-83. doi: 10.1001/archinternmed.2012.1993. PMID 22710744
- [Background] Dykstra PA. Older adult loneliness: myths and realities. Eur J Ageing. 2009 Jun;6(2):91-100. doi: 10.1007/s10433-009-0110-3. Epub 2009 Apr 4. PMID 19517025
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] McPherson, M., L. Smith-Lovin, and M.E. Brashears, Social isolation in America: Changes in core discussion networks over two decades. American sociological review, 2006. 71(3): p. 353-375.
- [Background] Steptoe A, Shankar A, Demakakos P, Wardle J. Social isolation, loneliness, and all-cause mortality in older men and women. Proc Natl Acad Sci U S A. 2013 Apr 9;110(15):5797-801. doi: 10.1073/pnas.1219686110. Epub 2013 Mar 25. PMID 23530191
- [Background] Taube E, Kristensson J, Sandberg M, Midlov P, Jakobsson U. Loneliness and health care consumption among older people. Scand J Caring Sci. 2015 Sep;29(3):435-43. doi: 10.1111/scs.12147. Epub 2014 May 14. PMID 24826811
- [Background] Gerst-Emerson K, Jayawardhana J. Loneliness as a public health issue: the impact of loneliness on health care utilization among older adults. Am J Public Health. 2015 May;105(5):1013-9. doi: 10.2105/AJPH.2014.302427. Epub 2015 Mar 19. PMID 25790413
- [Background] MacIntyre I, Corradetti P, Roberts J, Browne G, Watt S, Lane A. Pilot study of a visitor volunteer programme for community elderly people receiving home health care. Health Soc Care Community. 1999 May;7(3):225-232. doi: 10.1046/j.1365-2524.1999.00178.x. PMID 11560637
- [Background] Wright L, Vance L, Sudduth C, Epps JB. The Impact of a Home-Delivered Meal Program on Nutritional Risk, Dietary Intake, Food Security, Loneliness, and Social Well-Being. J Nutr Gerontol Geriatr. 2015;34(2):218-27. doi: 10.1080/21551197.2015.1022681. PMID 26106989
- [Background] Cattan M, Kime N, Bagnall AM. The use of telephone befriending in low level support for socially isolated older people--an evaluation. Health Soc Care Community. 2011 Mar;19(2):198-206. doi: 10.1111/j.1365-2524.2010.00967.x. Epub 2010 Nov 29. PMID 21114564

DOCUMENTS (2):
  • Study Protocol (2018-05-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03552328/Prot_000.pdf
  • Informed Consent Form (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03552328/ICF_001.pdf